CLINICAL TRIAL: NCT03431896
Title: Monitoring of Early Disease Progression in Hereditary Transthyretin Amyloidosis
Acronym: MED-hATTR
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1301
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Amyloidosis; Amyloid; Amyloid Neuropathies, Familial; Amyloid Cardiomyopathy; Amyloid - Primary; Transthyretin Amyloidosis; AL Amyloidosis
MeSH Terms: conditions — Amyloidosis; Alzheimer Disease; Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary: 1.) To evaluate the relative amount of misfolded ATTR oligomers in asymptomatic ATTR amyloid genetic carriers and correlate their levels with clinical symptoms and outcomes.
  1. Determine if misfolded ATTR oligomers are elevated compared to healthy control data obtained by Scripps during probe development
  2. Describe the levels longitudinally
  3. Determine if treatment with ATTR-specific medications (examples: diflunisal, doxycycline, ursodiol, tauroursodeoxycholic acid (TUDCA), green tea extract, curcumin, tafamidis, inotersen, patisiran) lead to reduction in the probe levels in those with elevated levels at baseline

SUMMARY:
This study measures circulating, misfolded ATTR oligomers in asymptomatic ATTRm amyloidosis genetic carriers longitudinally over five years.

DETAILED DESCRIPTION:
Recent advances in genetic testing have allowed for pathogenic mutation identification in family members of affected individuals prior to onset of symptoms. While the presence of mutation and the corresponding TTR kinetic stability have been directly linked to disease development, the molecular drivers of tissue specific degeneration have not been defined. We hypothesize that soluble misfolded TTR oligomer species may be circulating within the blood of these patients possibly years prior to amyloid deposition and could serve as an early biomarker and/or driver for disease development. In this line, The Scripps Research Institute has developed a peptide-based probe that specifically labels and integrates into misfolded TTR oligomers allowing the relative circulating concentration in the bloodstream to be determined. Longitudinal monitoring of untreated, asymptomatic TTR amyloid genetic carriers utilizing the Scripps probe is likely to provide novel insight into early disease progression. We also plan to utilize the Scripps probe to monitor disease progression in TTR amyloid genetic carriers currently undergoing treatment by observing how treatments affect the circulating misfolded TTR oligomers. Through enhanced understanding of early disease progression and treatment efficacy, our hope is to limit amyloid accumulation in cardiac and nerve tissue and delay the development of the invariably fatal TTR amyloid cardiomyopathy/neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known hereditary ATTR amyloidosis genetic mutations as identified by genetic testing.

Exclusion Criteria:

* Patients with ATTR amyloidosis identified as wild-type.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified through clinical practice and from Amyloid support groups
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average % change in oligomers in patients with new onset TTR amyloid symptoms | Annually over 5 years
  Change (%) for oligomer level at the time of TTR amyloid symptoms compared to baseline

SECONDARY OUTCOMES:
% change of oligomer levels relative to baseline level in patients with ATTR specific medication changes | Annually over 5 years
  Change (%) for oligomer level at the time of ATTR specific medication changes compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mazen A Hanna, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States